CLINICAL TRIAL: NCT07247188
Title: A Phase 3, Randomized, Modified Double-blind, Active-controlled, Parallel-group, 2-arm Study to Investigate the Safety and Immunogenicity of a Single Dose of a 21-valent Pneumococcal Conjugate Vaccine in Children and Adolescents With Sickle Cell Disease
Brief Title: Study of a Single Dose of a 21-valent Pneumococcal Conjugate Vaccine in Children and Adolescents With Sickle Cell Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PSK00026; U1111-1319-0153 (Other: WHO ICTRP)
Record Dates: First submitted 2025-11-19; First posted 2025-11-25 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Pneumococcal Vaccine; Pneumococcal Conjugate Vaccine
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Control method: Active-controlled
Who Masked: Participant
Masking Description: Modified double-blind:
  * Blinding for vaccine group assignment: participants and participant's parent(s)/legally acceptable representative(s), outcome assessors, Investigators, laboratory personnel, and Sponsor study staff
  * No blinding for vaccine group assignment: study staff preparing and administering the study interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigated Vaccine: PCV21 (Experimental): Participants will receive 1 intramuscular injection of the pneumococcal vaccine
  Interventions: Biological: PCV21
- Comparator Vaccine: 20vPCV (Active Comparator): Participants will receive 1 intramuscular injection of the pneumococcal vaccine
  Interventions: Biological: 20vPCV

INTERVENTIONS:
Biological: PCV21 — Investigational pneumococcal conjugate vaccine
  Arms: Investigated Vaccine: PCV21
Biological: 20vPCV — 20-valent pneumococcal conjugate vaccine
  Other Names: Prevnar 20
  Arms: Comparator Vaccine: 20vPCV

SUMMARY:
The purpose of this study is to measure whether PCV21 vaccine (investigational pneumococcal vaccine) is safe and can help the body to develop germ-fighting agents called "antibodies" (immunogenicity) compared with 20vPCV (licensed pneumococcal vaccine) when given as a single dose to children aged 2 to 17 years with sickle cell disease who had received or not a previous vaccination with pneumococcal conjugate or pneumococcal polysaccharide vaccine.

DETAILED DESCRIPTION:
The study duration per participant will be up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

AGE

* Aged 2 to 17 years on the day of inclusion.

TYPE OF PARTICIPANT AND DISEASE CHARACTERISTICS

* Participants who have a documented diagnosis of sickle cell disease (SCD) in their medical record.

SEX, CONTRACEPTIVE/BARRIER METHOD AND PREGNANCY TESTING REQUIREMENTS

* A participant is eligible to participate if the participant is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be pre-menarchal or surgically sterile. OR
  * Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 4 weeks after study intervention administration. A participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) within 25 hours before the study intervention.

INFORMED CONSENT

* Assent form has been signed and dated by the participant (based on local regulations), and, if applicable, informed consent form has been signed and dated by the parent(s) or another legally acceptable representative (LAR) and by an independent witness, if required by local regulations.

OTHER INCLUSIONS

* Participant and parent(s)/LAR are able to attend all scheduled visits and to comply with all study procedures.

Exclusion Criteria:

MEDICAL CONDITIONS

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy.
* History of microbiologically confirmed S. pneumoniae infection or disease.
* History of seizure or significant stable or progressive neurological disorders such as inflammatory nervous system diseases, encephalopathy, and cerebral palsy.
* Known systemic hypersensitivity to any of the study interventions components, or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances.
* Laboratory-confirmed thrombocytopenia, or known thrombocytopenia, as reported by the parent/LAR, contraindicating intramuscular (IM) injection.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM injection.
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.

For children/adolescents (6 to 17 YoA) only

* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion.

PRIOR/CONCOMITANT THERAPY

* Receipt of at least one dose of 20vPCV.
* For children aged < 6 years: receipt of < 3 doses of pneumococcal conjugate vaccine or any dose of 23-valent pneumococcal polysaccharide vaccine (PPSV23).
* For children and adolescents aged ≥ 6 years: receipt of PPSV23 < 5 years before study vaccination or last PCV dose < 8 weeks before study vaccination.
* Receipt of any vaccine in the 4 weeks preceding the study intervention administration or planned receipt of any vaccine in the 4 weeks following the study intervention administration, except for US licensed influenza vaccination, which may be received at least 2 weeks before or 2 weeks after study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines, as applicable per local recommendations.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Receipt of an oral or injectable antibiotic therapy for any acute illness within 72 hours prior to the first blood draw.

PRIOR/CONCURRENT CLINICAL STUDY EXPERIENCE

* Participation at the time of study enrollment (or in the 6 weeks preceding the first study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.

OTHER EXCLUSIONS For children (2 to 5 YoA) only

* Being in an emergency setting.
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study.

For children/adolescents (6 to 17 YoA) only

* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-01-07 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting immediate adverse events (AEs) | Within 30 minutes post-vaccination
  Unsolicited (spontaneously reported) systemic AEs after injection of a pneumococcal vaccine
Number of participants reporting solicited injection site and solicited systemic reactions | Up to Day 7 post-vaccination
Number of participants reporting unsolicited (spontaneously reported) injection site reactions and unsolicited systemic AEs after injection of a pneumococcal vaccine | Within 30 days post-vaccination
Number of participants reporting serious adverse events (SAEs) and adverse events of special interest (AESIs) | From day 0 to day 181
  SAEs and AESIs are collected throughout the study period
Number of participants with serotype-specific immunoglobulin G (IgG) concentrations for all serotypes included in PCV21 | On day 30 post-vaccination
  Ab (antibody) concentrations for each pneumococcal serotype measured by electro-chemiluminescence (ECL) assay

SECONDARY OUTCOMES:
Number of participants with serotype-specific IgG concentrations for all serotypes included in PCV21 | Pre-vaccination and at 30 days post-vaccination
  Ab concentrations for each pneumococcal serotype are measured by ECL assay
Number of participants with serotype specific opsonophagocytic activity (OPA) titers for all serotypes included in PCV21 | On day 30
  Serotype specific OPA titers for each pneumococcal serotype are determined by multiplex opsonophagocytic killing assay (MOPA)
Number of participants with serotype specific opsonophagocytic activity (OPA) titers for all serotypes included in PCV21 | Pre-vaccination and at 30 days post-vaccination
  Serotype specific OPA titers for each pneumococcal serotype are determined by multiplex opsonophagocytic killing assay (MOPA)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations Study Director, Study Director — Sanofi
Locations (1):
- Site # 8400006, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org